CLINICAL TRIAL: NCT01357551
Title: Maintenance After Initiation of Nutrition TrAINing (MAINTAIN)
Brief Title: Maintenance After Initiation of Nutrition TrAINing
Acronym: MAINTAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 11-040
Record Dates: First submitted 2011-05-13; First posted 2011-05-20 (Estimated); Results first posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-09

CONDITIONS: Obesity
Keywords: obesity; intervention studies; patient adherence
MeSH Terms: conditions — Obesity; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maintenance intervention (Experimental): Participants receive a theoretically-informed maintenance intervention for 42 weeks, followed by 14 weeks of no intervention contact to examine sustainability. The maintenance intervention involves in-person group visits that transition to individualized telephone calls, and the frequency of contact gradually decreases over time.
  Interventions: Behavioral: Maintenance intervention
- Usual care (No Intervention): Participants receive usual care for 56 weeks

INTERVENTIONS:
Behavioral: Maintenance intervention — Theoretically-informed maintenance intervention that involves in-person group visits that transition to individualized telephone calls, and the frequency of contact gradually decreases over time.
  Arms: Maintenance intervention

SUMMARY:
Obesity is the second leading cause of preventable deaths in the United States and is associated with a wide range of diseases. In people who are obese, weight loss improves blood pressure, dyslipidemia, glycemia, and arthritis symptoms; reduces medication use for several disease processes; increases physical functioning; and enhances health-related quality of life. The current study evaluated a theoretically informed maintenance intervention. If effective, this intervention could reduce the need for future clinic visits to treat obesity and its many associated illnesses.

DETAILED DESCRIPTION:
Obesity is the second leading cause of preventable deaths in the United States and is associated with a wide range of diseases. In people who are obese, weight loss improves blood pressure, dyslipidemia, glycemia, and arthritis symptoms; reduces medication use for several disease processes; increases physical functioning; and enhances health-related quality of life. Despite these benefits, most patients who achieve weight loss regain much of this weight within a year, and few effective behavioral weight maintenance interventions have been identified. Thus, there is a dire need for effective interventions that can promote weight loss maintenance. Theoretical and empirical studies indicate that behavior maintenance is a distinct state that involves different psychological processes and behavioral skills than initial behavior change. The few trials that have tested weight loss maintenance interventions have not taken this distinction into account, which may partially explain their modest findings. The current study evaluated the efficacy of a theoretically informed maintenance intervention compared to usual care. If efficacious, this intervention could reduce the need for future clinic visits to treat obesity and its many associated illnesses and could serve as a model for redesigning the MOVE! program. This 3.5-year study involved a two-arm, randomized, controlled trial. During the run-in phase, Veterans with BMI 30 kg/m2 participated in a 4-month, intensive, group-based weight loss program. Participants who lost at least 4 kg by the end of 4 months (n=222) were randomized to receive (a) usual care (n=112) for 56 weeks or (b) a theoretically-informed maintenance intervention (n=110) for 42 weeks months, followed by 14 weeks of no intervention contact to examine sustainability. The maintenance intervention involved in-person group visits that transition to individualized telephone calls, and the frequency of contact with the interventionist gradually tapered over time. Outcomes were assessed at randomization and at weeks 14, 26, 42, and 56 post-randomization. The hypotheses are that the maintenance intervention will result in at least 3.5 kg greater weight loss and greater improvements in caloric intake and physical activity over the study period, and that it will be cost-effective, compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* BMI >= 30 kg/m2
* Desire to lose weight
* Agrees to attend regular visits per study protocol
* Has a provider at the Durham Veterans Affairs Medical Center

Exclusion Criteria:

* Age >= 75 years old,
* Most recent serum creatinine >2.0 mg/dL in men, >1.7 mg/dL in women),
* Liver disease (cirrhosis, jaundice, or other stigmata of advanced liver disease),
* Type 1 diabetes,
* Hemoglobin A1c >= 12% in past 6 months
* unstable angina or coronary ischemia workup in past 3 months
* Female: pregnancy, breastfeeding, or lack of birth control if premenopausal
* Transplant recipient
* Pacemaker or defibrillator (bioelectric impedance assessment might interfere with these)
* Average systolic blood pressure in the past year >= 160 mmHg AND most recent BP >=160 mmHg
* Dementia, severe psychiatric illness (e.g., major depression), alcohol problem, or illicit substance abuse
* Weight loss of at least 10 lb in previous 3 months
* Enrollment in a weight loss program
* Unable to stand for study measurements
* history of weight loss surgery
* cancer not in remission
* current use of appetite suppressants or weight loss medication
* lack of reliable transportation or telephone

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2012-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corrine I Voils, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

REFERENCES:
- [Result] Voils CI, Gierisch JM, Yancy WS Jr, Sandelowski M, Smith R, Bolton J, Strauss JL. Differentiating Behavior Initiation and Maintenance: Theoretical Framework and Proof of Concept. Health Educ Behav. 2014 Jun;41(3):325-36. doi: 10.1177/1090198113515242. Epub 2013 Dec 16. PMID 24347145
- [Result] Voils CI, Gierisch JM, Olsen MK, Maciejewski ML, Grubber J, McVay MA, Strauss JL, Bolton J, Gaillard L, Strawbridge E, Yancy WS Jr. Study design and protocol for a theory-based behavioral intervention focusing on maintenance of weight loss: the Maintenance After Initiation of Nutrition TrAINing (MAINTAIN) study. Contemp Clin Trials. 2014 Sep;39(1):95-105. doi: 10.1016/j.cct.2014.08.002. Epub 2014 Aug 10. PMID 25117805
- [Derived] Gavin KL, Almeida EJ, Voils CI, Crane MM, Shaw R, Yancy WS Jr, Pendergast J, Olsen MK. Comparison of weight captured via electronic health record and cellular scales to the gold-standard clinical method. Obes Sci Pract. 2023 Jan 12;9(4):337-345. doi: 10.1002/osp4.656. eCollection 2023 Aug. PMID 37546286
- [Derived] Funk LM, Grubber JM, McVay MA, Olsen MK, Yancy WS, Voils CI. Patient predictors of weight loss following a behavioral weight management intervention among US Veterans with severe obesity. Eat Weight Disord. 2018 Oct;23(5):587-595. doi: 10.1007/s40519-017-0425-6. Epub 2017 Aug 29. PMID 28853051
- [Derived] Voils CI, Olsen MK, Gierisch JM, McVay MA, Grubber JM, Gaillard L, Bolton J, Maciejewski ML, Strawbridge E, Yancy WS Jr. Maintenance of Weight Loss After Initiation of Nutrition Training: A Randomized Trial. Ann Intern Med. 2017 Apr 4;166(7):463-471. doi: 10.7326/M16-2160. Epub 2017 Feb 21. PMID 28241185

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 573 people were consented. Of those, 69 did not return to provide a weight at study entry. Of the 504 who provided a weight at study entry, 200 dropped out, 82 lost < 4 kg, and 222 lost at least 4 kg and thus were eligible for randomization in the maintenance phase.
Groups:
- Maintenance Intervention: Participants receive theoretically-informed maintenance intervention for 42 weeks, followed by 16 weeks of no intervention contact to examine sustainability.
  Interventions: Theoretically-informed maintenance intervention that involves in-person group visits that transition to individualized telephone calls, and the frequency of contact with the interventionist gradually decreases over time.
Period: Overall Study
Arm/Group | Maintenance Intervention | Usual Care
Started | 110 | 112
Completed | 88 | 101
Not Completed | 22 | 11
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 16 | 6

BASELINE CHARACTERISTICS:
Groups:
- Maintenance Intervention: Participants are randomized to a theoretically-informed maintenance intervention for 42 weeks, followed by 14 weeks of no intervention contact to examine sustainability. The maintenance intervention will involve in-person group visits that transition to individualized telephone calls, and the frequency of contact with the interventionist will gradually taper over time.
  Interventions: Theoretically-informed maintenance intervention that involves in-person group visits that transition to individualized telephone calls, and the frequency of contact with the interventionist will gradually taper over time.
- Usual Care: Participants are randomized to receive usual care for 56 weeks
- Total: Total of all reporting groups
Arm/Group | Maintenance Intervention | Usual Care | Total
Number analyzed (Participants) | 110 | 112 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (8.3) | 62.0 (8.3) | 61.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 93 | 95 | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 105 | 111 | 216
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 38 | 45 | 83
  White | 67 | 62 | 129
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 110 | 112 | 222
Weight loss during initiation phase [Mean (Standard Deviation); unit: kilograms] | 7.2 (2.8) | 7.2 (3.4) | 7.2 (3.1)
Weight [Mean (Standard Deviation); unit: kilograms] | 102.1 (19.8) | 105.0 (21.0) | 103.6 (20.4)
Body mass index [Mean (Standard Deviation); unit: kilograms per meter squared] | 33.3 (5.7) | 34.6 (6.4) | 34.0 (6.1)
Education [Number; unit: participants]
  high school graduate | 106 | 111 | 217
  not high school graduate | 3 | 1 | 4
  missing | 1 | 0 | 1
Current tobacco user [Number; unit: participants]
  yes | 5 | 9 | 14
  no | 105 | 102 | 207
  missing | 0 | 1 | 1
Employment status [Number; unit: participants]
  working full time or part-time | 33 | 28 | 61
  retired | 59 | 65 | 124
  other/disabled | 17 | 18 | 35
  missing | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Weight
Time Frame: 56 weeks post-randomization
Measure: Mean (Standard Deviation); unit: kilograms
Groups:
- Maintenance Intervention: Participants are randomized to a theoretically-informed maintenance intervention for 42 weeks, followed by 16 weeks of no intervention contact to examine sustainability. The maintenance intervention will involve in-person group visits that transition to individualized telephone calls, and the frequency of contact with the interventionist will gradually taper over time.
  Interventions: Theoretically-informed maintenance intervention that involves in-person group visits that transition to individualized telephone calls, and the frequency of contact with the interventionist will gradually taper over time.
Arm/Group | Maintenance Intervention | Usual Care
Number analyzed (Participants) | 110 | 112
kilograms | 99.2 (17.7) | 105.7 (20.1)
Statistical Analysis 1: Comparison: Maintenance Intervention vs Usual Care; The sample size estimate was based on the primary hypothesis that patients randomized to receive the maintenance intervention would have less mean weight regain at week 56 than those randomized to usual care. The week 0 standard deviation was estimated as 24.6kg, the correlation between week 0 and week 56 as 0.95, and the week 56 dropout rate as 10%. To detect a difference of 3.5 kg with 90% power and a type I error rate of 5%, 230 total (115 in each group) randomized patients were needed; Test type: Superiority or Other; p = .04, Mixed Models Analysis — A priori threshold was p<.05; Parameters included common intercept, initial weight loss stratum, dummy-coded time, and indicators for the maintenance X each follow-up time point; Mean Difference (Final Values) = 1.61, 95% CI 2-sided [.07 to 3.13], Standard Error of Mean .78

2. Secondary Outcome: Estimated Daily Caloric Intake
Description: Based on self-report using Block Brief Food Frequency Questionnaire
Time Frame: 56 weeks
Measure: Mean (Standard Deviation); unit: kcal per day
Groups:
- Maintenance Intervention: Participants receive a theoretically-informed maintenance intervention for 42 weeks, followed by 16 weeks of no intervention contact to examine sustainability. The maintenance intervention involves in-person group visits that transition to individualized telephone calls, and the frequency of contact gradually decreases over time.
  Interventions: Theoretically-informed maintenance intervention that involves in-person group visits that transition to individualized telephone calls, and the frequency of contact gradually decreases over time.
Arm/Group | Maintenance Intervention | Usual Care
Number analyzed (Participants) | 110 | 112
kcal per day | 1207.5 (548.3) | 1339.1 (750.5)
Statistical Analysis 1: Comparison: Maintenance Intervention vs Usual Care; The hypothesis was that patients randomized to receive the maintenance intervention would have less caloric intake at week 56 than those randomized to usual care; Test type: Superiority or Other; p = .11, Mixed Models Analysis; Common intercept, initial weight loss stratum, indicators for week 26 & 56, group X time interaction; Mean Difference (Net) = -125.49, 95% CI 2-sided [-280.71 to 29.72], Standard Error of Mean 78.64

3. Secondary Outcome: Estimated Metabolic Minutes of Walking Per Week
Description: self-reported based on short form of International Physical Activity Questionnaire
Time Frame: 56 weeks
Measure: Mean (Standard Deviation); unit: metabolic minutes per week
Arm/Group | Maintenance Intervention | Usual Care
Number analyzed (Participants) | 110 | 112
metabolic minutes per week | 680.72 (721.23) | 665.43 (822.30)
Statistical Analysis 1: Comparison: Maintenance Intervention vs Usual Care; The hypothesis was that patients randomized to receive the maintenance intervention would have higher rates of walking per week at week 56 than those randomized to usual care; Test type: Superiority or Other; p = .91, Mixed Models Analysis; Common intercept, initial weight loss stratum, indicators for week 26 & 56, group X time interaction; negative binomial distribution with log link; incidence rate ratio = 1.03, 95% CI 2-sided [0.63 to 1.68], Standard Error of Mean .26

4. Secondary Outcome: Estimated Metabolic Minutes of Moderate Physical Activity Per Week
Description: self-reported based on short form of International Physical Activity Questionnaire
Time Frame: 56 weeks
Measure: Mean (Standard Deviation); unit: metabolic minutes per week
Arm/Group | Maintenance Intervention | Usual Care
Number analyzed (Participants) | 110 | 112
metabolic minutes per week | 783.40 (1175.57) | 810.25 (1215.14)
Statistical Analysis 1: Comparison: Maintenance Intervention vs Usual Care; The hypothesis was that patients randomized to receive the maintenance intervention would have higher rates of moderate physical activity per week at week 56 than those randomized to usual care; Test type: Superiority or Other; p = .83, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; incidence rate ratio = 1.07, 95% CI 2-sided [0.57 to 2.03], Standard Error of Mean .35

ADVERSE EVENTS:
Time Frame: 56-week study period
Groups:
- Maintenance Intervention: Participants receive a theoretically-informed maintenance intervention for 42 weeks, followed by 16 weeks of no intervention contact to examine sustainability. The maintenance intervention involves in-person group visits that transition to individualized telephone calls, and the frequency of contact gradually decreases over time.
  Maintenance intervention: Theoretically-informed maintenance intervention that involves in-person group visits that transition to individualized telephone calls, and the frequency of contact gradually decreases over time.
Arm/Group | Maintenance Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 4/110 | 1/112
Other Adverse Events (participants affected / at risk) | 0/110 | 0/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maintenance Intervention (N=110) | Usual Care (N=112)
Emergency room visit due to high blood pressure (Cardiac disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1)
emergency room visit due to knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Emergency room visit due to anxiety (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
May not generalize to other populations; relatively short length of follow-up; use of self-reported secondary outcome measures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes